CLINICAL TRIAL: NCT06317831
Title: LetS Get fUnctional! FuNctional Status in pEople With intersTitial Lung Disease - the SUNSET Study
Brief Title: LetS Get fUnctional! FuNctional Status in pEople With intersTitial Lung Disease
Acronym: SUNSET
Status: Recruiting | Type: Observational
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Other Study IDs: 2023.03936.BDANA
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Interstitial Lung Diseases
Keywords: Functional Status; Interstitial lung diseases; Assessment; Patient-centered care
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to i) To characterize the functional status and explore the determinants of functional status decline of people with IlD ii)To determine the measurement properties of functional status instruments in people with Interstitial lung diseases (ILD) iii) To identify the impact of ILD and the participants' perspectives on functional status through interviews iv) Explore the progression of functional status progression in people with ILD and v) Develop a multidimensional index, incorporating functional status parameters, to predict mortality in people with ILD.

Patients with ILD will be recruited via the pulmonology services at hospitals, namely from Centro Hospitalar de Vila Nova de Gaia/Espinho (CHVNG/E), Centro Hospitalar do Baixo Vouga (CHBV) and Centro Hospitalar de Entre o Douro e Vouga (CHEDV). Sociodemographic, clinical characteristics (i.e., smoking habits, vital signs and symptoms), anthropometric (i.e., height and weight to compute body mass index) and general clinical data (i.e., medication, oxygen therapy, non-invasive ventilation, acute exacerbations, hospitalizations and number of hospital admissions in the last month and year, length of stay), as well as prior and follow-up spirometric measurements and arterial blood gas will be collected from clinical records for patients' characterization. Mortality and rehospitalizations will be explored during the study period. Peripheral muscle strength, functional status, daily physical activity, self-reported symptoms, functional status, impact of the disease and health-related quality of life. Qualitative data from interviews.

The assessments will be conducted at 6 time points: baseline and 1 week after for instrument validation, followed by assessments every 6 months for 2 years.

It is expected that: i) Functional status limitations can be comprehensively identified and measured in individuals with ILD. ii) Some measures are valid and reliable indicators of functional status in individuals with ILD. iii) Different profiles of functional status progression will be identified in individuals with ILD, including stable, slow, and fast decline. iv) A multidimensional index incorporating functional status will improve the accuracy of predicting mortality and outperform the predictive ability of the current GAP Index.

DETAILED DESCRIPTION:
Functional status is a fundamental, patient-centred and multidimensional outcome for individuals with interstitial lung disease (ILD). Functional status decline is the most frequent impact reported in this population. It is often associated with an increased dependency on others, loss of productivity and premature death. It is also an important predictor of exacerbations, hospitalisations, readmissions, and mortality. Functional status decline is so overwhelming for individuals and society, that it has been recently recognised as an international top priority for patient-centred research in ILD. Yet, little is known how functional status is impaired and progresses in ILD, limiting the help health professionals are able to provide to optimise care.

ILD are a highly disabling group of chronic respiratory diseases characterised by widespread inflammation and scarring (fibrosis) of the lung. In people with ILD, the destruction of the pulmonary capillary bed and vasoconstriction, results in impaired gas exchange and circulatory limitation, which can lead to reduced exercise capacity. Exercise capacity may be further limited due to peripheral muscle dysfunction caused by physical deconditioning and drug-induced myopathy from ILD treatment with corticosteroids. Taken together these factors contribute to the high symptom burden experienced. This population, therefore, presents pulmonary (e.g., dyspnoea, cough) and extra-pulmonary (e.g., decreased exercise tolerance, skeletal muscle dysfunction, fatigue) traits and experience a downward spiral of debilitating symptoms and functional status decline.

Functional status is defined as the ability to perform normal daily activities required to meet basic needs, fulfil usual roles, and maintain health and well-being. It includes functional capacity, i.e., an individual's maximum capacity to perform daily life activities in a standardized environment; and functional performance, i.e., activities people actually do during the course of their daily life. Adequate assessment of functional status must, therefore, include measures of functional capacity and performance, to identify the presence or absence of decline and inform on preventive and/or rehabilitative strategies. Studies focussing on the comprehensive assessment of functional status in people with ILD using reliable and validated instruments are, however, lacking.

Therefore, the primary aim of SUNSET study is to characterize the functional status and explore the determinants of functional status decline of people with ILD.

Secondary aims are to: i) To determine the measurement properties of functional status instruments in people with ILD ii) To identify the impact of ILD and the participants' perspectives on functional status through interviews iii) Explore the progression of functional status progression in people with ILD and iv) Develop a multidimensional index, incorporating functional status parameters, to predict mortality in people with ILD.

According to the COnsensus-based Standards for the selection of health Measurement INstruments (COSMIN) guideline, a minimum sample size of 100 will be required for task 1.

For task 2, number of participants needed for interviews will be determined by data saturation.

For task 3, a sample size estimation was performed in GPower to detect a small effect size (eta^2=0.02), with 80% power, 5% significance level and moderate correlation among repeated measures (r=0.5) in a repeated measures analysis of variance. The minimum sample size estimation was 81 participants Considering a dropout rate of 50%, we will aim to recruit 122 participants.

This study is a multicentric observational longitudinal research project comprising four tasks. It involves collaboration between institutions, namely the University of Aveiro, along with three healthcare facilities: Centro Hospitalar de Vila Nova de Gaia/Espinho (CHVNG/E), Centro Hospitalar do Baixo Vouga (CHBV), and Centro Hospitalar de Entre o Douro e Vouga (CHEDV). Task 1 aims to validate the measures of functional status. For this, two assessment moments will be performed. The first assessment will be conducted at baseline and will be in line with the routine appointment. The second assessment will be conducted 7 days after baseline. Task 2 will use the information collected in Task 1 and conduct semi-structured individual interviews to characterize the functional status from the perspective of people with ILD. Task 3 will then conduct an observational longitudinal study using the most valid and reliable measures of functional status identified in task 1 and mortality rates will be explored during task 3. For this, patients will be contacted to participate in four timepoints of assessment (at 6, 12, 18, and 24 months) which will be in line with the routine appointment. Table 1 details the measurements performed in each timepoint. If an outcome measure is found to not be valid and reliable during task 1, that outcome measure will not be collected in task 3 nor replaced by another outcome measure. In Task 4, the data collected in Task 3 will be used to develop a multidimensional index incorporating functional status parameters to predict mortality in people with ILD. The study assessments will take approximately 90 minutes and will take place at Centro Hospitalar de Vila Nova de Gaia/Espinho (CHVNG/E), Centro Hospitalar do Baixo Vouga (CHBV), and Centro Hospitalar de Entre o Douro e Vouga (CHEDV).

Patients with ILD will be recruited via the pulmonology services at hospitals. Pulmonologists will explain the study briefly and inform the researchers about interested participants. The researchers will provide further information about the study, clarify any doubts and collect the informed consent. Participants will be eligible if they are: i) ≥18 years, ii) diagnosed with any type of ILD, iii) fluent in Portuguese and iv) able to provide informed consent. Participants will be excluded if they have: i) other respiratory diseases ii) a history of acute cardiac/respiratory condition in the previous month; iii) present signs of cognitive impairment; iv) significant cardiovascular, neurological and/or musculoskeletal disease that may limit their participation; v) current neoplasia, vi) other autoimmune diseases (aside from ILD). Once task 1 is finished, included participants will be contacted again to verify if they still match the inclusion/exclusion criteria and are still willing to participate in task 3.

Baseline data will be collected: Sociodemographic, clinical characteristics (i.e., smoking habits, vital signs and symptoms), anthropometric (i.e., height and weight to compute body mass index) and general clinical data (i.e., medication, oxygen therapy, non-invasive ventilation, acute exacerbations, hospitalizations and number of hospital admissions in the last month and year, length of stay), as well as prior and follow-up lung function and arterial blood gas will be collected from clinical records for patients' characterization. Mortality and rehospitalizations will be explored during the study period. Peripheral muscle strength, functional status, daily physical activity, self-reported symptoms, functional status, impact of the disease and health-related quality of life. Qualitative data from interviews.

Data analysis will be conducted using the Statistical Package for the Social Sciences (SPSS) software, incorporating both descriptive and inferential statistics. To examine changes in outcome measures, data from baseline and subsequent assessments will be compared. Additionally, the interviews will be transcribed and analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Diagnosed with any type of ILD
* Fluent in Portuguese
* Able to provide informed consent.

Exclusion Criteria:

* Other respiratory diseases
* A history of acute cardiac/respiratory condition in the previous month
* Present signs of cognitive impairment
* Significant cardiovascular, neurological and/or musculoskeletal disease that may limit their participation
* Current neoplasia
* Other autoimmune diseases (aside from ID).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Interstitial Lung Disease
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Short physical performance battery (SPPB) | Two measurements will be assessed at baseline and one at each follow-up (baseline, 6 months, 12 months, 18 months and 24 months)
  Patients' functional level will be assessed with the short physical performance battery, a simple and easy to perform tool that includes the four-meter gait speed test, the five-repetition sit-to-stand test and a balance test, and gives a total score based on the performance in each of those tests.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | Only one measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months).
  The Six Minute Walk Test is the gold standard exercise test and has been validated in people with ILD and is commonly used to assess functional status. The 6MWD is valid and reliable measure in people with ILD, with excellent intra-class correlation coefficients (ICCs= 0.82-0.99).
The 1-minute sit-to-stand | Two measurements will be assessed at baseline and one at each follow-up (baseline, 6 months, 12 months, 18 months and 24 months)
  The 1-minute sit-to-stand test will be used to also assess functional status.
The grocery shelving task | Two measurements will be conducted in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months) due to the presence of a learning effect with this test.
  The grocery shelving task is valid, reliable and responsive functional outcome measure that incorporates unsupported arm activity in patients with chronic respiratory disease.
The Physical Performance Test (PPT) | Two measurements will be assessed at baseline and one at each follow-up (baseline, 6 months, 12 months, 18 months and 24 months)
  The Physical Performance Test (PPT) is valid and reliable established measure of physical function status.
Handgrip strenght | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Participants' isometric handgrip muscle strength will be evaluated using a hydraulic hand dynamometer and measured in kilograms.
Peripheral muscle strength | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months).
  Participants' isometric biceps and quadriceps muscle strength will be collected with a hand-held dynamometer and measured in kilogram-force.
The Tilburg Frailty Indicator (TFI) | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The Tilburg Frailty Indicator (TFI) is a self-report user-friendly questionnaire for assessing multidimensional frailty among community-dwelling older people and has been used in people with chronic obstructive pulmonary disease. TFI is valid and reliable instrument to assess frailty.
The Canadian Occupational Performance Measure (COPM) | Three measurements will be assessed at baseline and one at each follow-up (baseline, 6 months, 12 months, 18 months and 24 months)
  The Canadian Occupational Performance Measure (COPM) is a reliable and responsive measure of a client's self-perception of occupational performance in the areas of self-care, productivity, and leisure. It has been used in chronic obstructive pulmonary disease.
Symptoms of fatigue | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The level of fatigue on a daily basis will be collected with the Checklist of Individual Strength 8 (CIS-8).
Symptoms of fatigue | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Patients' self-reported level of fatigue will be collected at rest, using the modified Borg scale.
Symptoms of dyspnoea | One measurement will be assessed in each timepoint (baselinre, 6 months, 12 months, 18 months and 24 months)
  Patients' self-reported level of dyspnoea will be collected at rest, using the modified Borg scale.
The Pulmonary Functional Status and Dyspnea Questionnaire Modified version (PFSDQ-M) | Three measurements will be assessed at baseline and one at each follow-up (baseline, 6 months, 12 months, 18 months and 24 months)
  The Pulmonary Functional Status and Dyspnea Questionnaire Modified version (PFSDQ-M) is a disease specific questionnaire with three domains: influence of dyspnea during activity of daily living (ADL), influence of fatigue on ADLs and change experienced by the patient in ADLs. Is valid and reliable questionnaire to assess ADL limitations in patients with COPD chronic obstructive pulmonary disease.
Health-related quality of life (HRQOL) | Only one measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The King's Brief Interstitial Lung Disease (K-BILD) will be used to evaluate health-related quality of life in individuals with interstitial lung disease
Health-related quality of life (HRQOL) | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The St George's Respiratory Questionnaire on Respiratory Pulmonary Fibrosis version (SGRQ-i), will be used to assess health-related quality of life in individuals with interstitial lung disease
London Chest Activities of Daily Living (LCADL) | Only one measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Patients' level of dyspnoea performing activities of daily living and functional status will be assessed with th London Chest Activities of Daily Living questionnaire.
Daily physical activity | Only one measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Physical activity will be objectively quantified, as an exploratory outcome, for managing the influence of physical activity on functional status assessment, with an Actigraph GT3X (Actigraph LLC Pensacola, FL, USA).
Qualitative data: Interviews | Only one measurement will be assessed at baseline (baseline, 6 months, 12 months, 18 months and 24 months)
  participants will be invited to take part in face-to-face, semi-structured individual interviews to understand the impact of ILD and participants' perspectives on functional status.
Number of hospitalizations | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Patients' number of hospitalizations in the previous year and during the follow-up period, as well as the length of stay for each hospitalization, will be assessed by asking the patient to self-report.
Acute exacerbations | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  Patients' number of acute exacerbations will be assessed by asking the patient to self-report.
Non-invasive ventilation | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The patients' use of non-invasive ventilation will be assessed by asking them to self-report.
Oxygen therapy | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The patients' use of oxygen therapy will be assessed by asking them to self-report.
Medication | One measurement will be assessed in each timepoint (baseline, 6 months, 12 months, 18 months and 24 months)
  The patients' medication will be assessed by asking them to self-report.
Mortality | One measurement will be assessed in each timepoint (6 months, 12 months, 18 months and 24 months)
  Patients who died after being included in the study will be identified by consulting the pneumologists.

OTHER OUTCOMES:
Weight | One measurement will be assessed in each timepoint (6 months, 12 months, 18 months and 24 months)
  The participants' weight will be assessed in kilograms.
Height | One measurement will be assessed in each timepoint (6 months, 12 months, 18 months and 24 months)
  The participants' weight will be assessed in meters.
Body mass index | One measurement will be assessed in each timepoint.
  Patients' body mass index will be assessed in kg/m^2 based on patients' height and weight.
Heart rate | One measurement will be assessed in each timepoint.
  Heart rate will be assessed in beats per minute using a oximeter and blood pressure meter.
Respiratory rate | One measurement will be assessed in each timepoint.
  Respiratory rate will be assessed by direct observation, counting the number of respiratory cycles.
Blood pressure | One measurement will be assessed in each timepoint.
  Blood pressure (systolic and diastolic) will be assessed using a blood pressure meter.
Peripheral Oxygen Saturation | The measurements will be collected before and after the six-minute walk test in each timepoint (6 months, 12 months, 18 months and 24 months)
  Peripheral oxygen saturation will be assessed with a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronson KI, Danoff SK, Russell AM, Ryerson CJ, Suzuki A, Wijsenbeek MS, Bajwah S, Bianchi P, Corte TJ, Lee JS, Lindell KO, Maher TM, Martinez FJ, Meek PM, Raghu G, Rouland G, Rudell R, Safford MM, Sheth JS, Swigris JJ. Patient-centered Outcomes Research in Interstitial Lung Disease: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2021 Jul 15;204(2):e3-e23. doi: 10.1164/rccm.202105-1193ST. PMID 34283696
- [Background] Hilberg O, Hoffmann-Vold AM, Smith V, Bouros D, Kilpelainen M, Guiot J, Morais A, Clemente S, Daniil Z, Papakosta D, Fretheim H, Neves S, Alfaro TM, Antoniou KM, Valveny N, Asijee G, Soulard S, Wuyts W. Epidemiology of interstitial lung diseases and their progressive-fibrosing behaviour in six European countries. ERJ Open Res. 2022 Jan 24;8(1):00597-2021. doi: 10.1183/23120541.00597-2021. eCollection 2022 Jan. PMID 35083316
- [Background] Dowman L, Hill CJ, May A, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2021 Feb 1;2(2):CD006322. doi: 10.1002/14651858.CD006322.pub4. PMID 34559419
- [Background] Tonelli R, Cocconcelli E, Lanini B, Romagnoli I, Florini F, Castaniere I, Andrisani D, Cerri S, Luppi F, Fantini R, Marchioni A, Beghe B, Gigliotti F, Clini EM. Effectiveness of pulmonary rehabilitation in patients with interstitial lung disease of different etiology: a multicenter prospective study. BMC Pulm Med. 2017 Oct 10;17(1):130. doi: 10.1186/s12890-017-0476-5. PMID 29017478
- [Background] Leidy NK. Functional status and the forward progress of merry-go-rounds: toward a coherent analytical framework. Nurs Res. 1994 Jul-Aug;43(4):196-202. PMID 8047422
- [Background] Kocks JW, Asijee GM, Tsiligianni IG, Kerstjens HA, van der Molen T. Functional status measurement in COPD: a review of available methods and their feasibility in primary care. Prim Care Respir J. 2011 Sep;20(3):269-75. doi: 10.4104/pcrj.2011.00031. PMID 21523316
- [Background] Dedding C, Cardol M, Eyssen IC, Dekker J, Beelen A. Validity of the Canadian Occupational Performance Measure: a client-centred outcome measurement. Clin Rehabil. 2004 Sep;18(6):660-7. doi: 10.1191/0269215504cr746oa. PMID 15473118
- [Background] Medina-Mirapeix F, Bernabeu-Mora R, Llamazares-Herran E, Sanchez-Martinez MP, Garcia-Vidal JA, Escolar-Reina P. Interobserver Reliability of Peripheral Muscle Strength Tests and Short Physical Performance Battery in Patients With Chronic Obstructive Pulmonary Disease: A Prospective Observational Study. Arch Phys Med Rehabil. 2016 Nov;97(11):2002-2005. doi: 10.1016/j.apmr.2016.05.004. Epub 2016 May 30. PMID 27255806
- [Background] Reuben DB, Siu AL. An objective measure of physical function of elderly outpatients. The Physical Performance Test. J Am Geriatr Soc. 1990 Oct;38(10):1105-12. doi: 10.1111/j.1532-5415.1990.tb01373.x. PMID 2229864
- [Background] Hill CJ, Denehy L, Holland AE, McDonald CF. Measurement of functional activity in chronic obstructive pulmonary disease: the grocery shelving task. J Cardiopulm Rehabil Prev. 2008 Nov-Dec;28(6):402-9. doi: 10.1097/HCR.0b013e31818c3c65. PMID 19008696
- [Background] Briand J, Behal H, Chenivesse C, Wemeau-Stervinou L, Wallaert B. The 1-minute sit-to-stand test to detect exercise-induced oxygen desaturation in patients with interstitial lung disease. Ther Adv Respir Dis. 2018 Jan-Dec;12:1753466618793028. doi: 10.1177/1753466618793028. PMID 30091679
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Dowman L, McDonald CF, Hill CJ, Lee A, Barker K, Boote C, Glaspole I, Goh N, Southcott A, Burge A, Ndongo R, Martin A, Holland AE. Reliability of the hand held dynamometer in measuring muscle strength in people with interstitial lung disease. Physiotherapy. 2016 Sep;102(3):249-55. doi: 10.1016/j.physio.2015.10.002. Epub 2015 Oct 22. PMID 26596172
- [Background] Karagiannis C, Savva C, Korakakis V, Matheou I, Adamide T, Georgiou A, Xanthos T. Test-Retest Reliability of Handgrip Strength in Patients with Chronic Obstructive Pulmonary Disease. COPD. 2020 Oct;17(5):568-574. doi: 10.1080/15412555.2020.1808604. Epub 2020 Aug 19. PMID 32814452
- [Background] Reilly CC, Bausewein C, Garrod R, Jolley CJ, Moxham J, Higginson IJ. Breathlessness during daily activity: The psychometric properties of the London Chest Activity of Daily Living Scale in patients with advanced disease and refractory breathlessness. Palliat Med. 2017 Oct;31(9):868-875. doi: 10.1177/0269216316680314. Epub 2016 Dec 15. PMID 27932629
- [Background] Zhang X, Tan SS, Bilajac L, Alhambra-Borras T, Garces-Ferrer J, Verma A, Koppelaar E, Markaki A, Mattace-Raso F, Franse CB, Raat H. Reliability and Validity of the Tilburg Frailty Indicator in 5 European Countries. J Am Med Dir Assoc. 2020 Jun;21(6):772-779.e6. doi: 10.1016/j.jamda.2020.03.019. Epub 2020 May 6. PMID 32387112
- [Background] Patel AS, Siegert RJ, Brignall K, Gordon P, Steer S, Desai SR, Maher TM, Renzoni EA, Wells AU, Higginson IJ, Birring SS. The development and validation of the King's Brief Interstitial Lung Disease (K-BILD) health status questionnaire. Thorax. 2012 Sep;67(9):804-10. doi: 10.1136/thoraxjnl-2012-201581. Epub 2012 May 3. PMID 22555278
- [Background] Van Remoortel H, Raste Y, Louvaris Z, Giavedoni S, Burtin C, Langer D, Wilson F, Rabinovich R, Vogiatzis I, Hopkinson NS, Troosters T; PROactive consortium. Validity of six activity monitors in chronic obstructive pulmonary disease: a comparison with indirect calorimetry. PLoS One. 2012;7(6):e39198. doi: 10.1371/journal.pone.0039198. Epub 2012 Jun 20. PMID 22745715
- [Background] Terwee CB, Prinsen CAC, Chiarotto A, Westerman MJ, Patrick DL, Alonso J, Bouter LM, de Vet HCW, Mokkink LB. COSMIN methodology for evaluating the content validity of patient-reported outcome measures: a Delphi study. Qual Life Res. 2018 May;27(5):1159-1170. doi: 10.1007/s11136-018-1829-0. Epub 2018 Mar 17. PMID 29550964
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585